CLINICAL TRIAL: NCT01828385
Title: Effect of Magnesium Sulfate on the Reversal of Neuromuscular Blockade With Sugammadex: a Prospective, Randomized Double-blind Trial
Brief Title: Effect of Magnesium on the Recovery Time of Neuromuscular Blockade With Sugammadex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Hospital Federal de Bonsucesso (Other)
Responsible Party: Principal Investigator, Paulo Alipio Germano Filho, MD, MSc, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAGF-01M
Record Dates: First submitted 2013-04-05; First posted 2013-04-10 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Neuromuscular Blockade
Keywords: Physiological Effects of Drugs; Rocuronium; Sugammadex sodium; Magnesium; Molecular Mechanisms of Pharmacological Action; Neuromuscular block, antagonism; Pharmacologic Actions
MeSH Terms: interventions — Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Mg (Experimental): Magnesium sulfate 40 mg.kg-1 + rocuronium 0.6 mg.kg-1 + sugammadex 2 mg.kg-1
  Interventions: Drug: Magnesium Sulfate
- Group C (Active Comparator): Saline 100 ml + rocuronium 0.6 mg.kg-1 + sugammadex 2 mg.kg-1
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Magnesium Sulfate — Magnesium sulfate + rocuronium + sugammadex
  Arms: Group Mg
Drug: Saline — Saline + rocuronium + sugammadex
  Arms: Group C

SUMMARY:
The aim of this study is to determine the recovery time of moderate neuromuscular blockade with sugammadex in adults pretreated with magnesium sulfate.

DETAILED DESCRIPTION:
Sugammadex is a novel neuromuscular blocking reversal agent. Its mechanism of action is the encapsulation of rocuronium and vecuronium molecules. Numerous studies show a potential role of magnesium in reducing anesthetic requirements, sympathetic response to surgical trauma, antinociceptive action and neuroprotective effects. However, its use is limited because magnesium potentiates non-depolarizing neuromuscular blocking agents.

Primary outcome: evaluate the effect of pretreatment with magnesium sulfate on the time reversal with sugammadex (recovery of the T4/T1 ratio = 0.9) of moderate neuromuscular blockade (two answers to a train-of-four TOF) induced by rocuronium.

Secondary outcome: evaluate severe respiratory events, the incidence of residual neuromuscular blockade in the post anesthesia recovery room and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* ASA physical status 1 or 2
* weight BMI 18.5-24.9
* otorhinolaryngological surgeries

Exclusion Criteria:

* major surgery associated with massive blood loss or fluid replacement
* any known allergy to magnesium sulphate or any other study drugs
* pregnant
* anatomical malformations expected to result in a difficult intubation;
* known or suspected neuromuscular disorders and/or significant hepatic or renal dysfunction
* administration of any medication known to interfere with neuromuscular blocking agents (such as anticonvulsants, aminoglycosides, calcium channel blockers and magnesium containing medications)
* hypomagnesemia, hypermagnesemia, hypocalcemia, hypercalcemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Recovery time of moderate neuromuscular blockade with sugammadex in adults pretreated with magnesium sulfate | 3 hours
  When T1 reached 25%, a single bolus dose of sugammadex 2 mg.kg-1 was administered to facilitate the recovery. The times to reach a TOF ratio of 0.9 and T1 height value were measured.

SECONDARY OUTCOMES:
Assess severe respiratory events, the incidence of residual neuromuscular blockade in anesthesia recovery room | 4 hours
  Clinical tests and contraction of the adductor pollicis muscle in response to ulnar nerve train-of-four (TOF) stimulation was acceleromyographically quantified using a TOF-Watch SX.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo A Germano Filho, MD, Principal Investigator — Hospital Federal de Bonsucesso; Núbia V Figueiredo, PhD, Study Director — Universidade Federal do Rio de Janeiro; Ismar L Cavalcanti, PhD, Study Director — Universidade Federal do Rio de Janeiro
Locations (1):
- Hospital Federal de Bonsucesso, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Herroeder S, Schonherr ME, De Hert SG, Hollmann MW. Magnesium--essentials for anesthesiologists. Anesthesiology. 2011 Apr;114(4):971-93. doi: 10.1097/ALN.0b013e318210483d. PMID 21364460
- [Background] Sauer M, Stahn A, Soltesz S, Noeldge-Schomburg G, Mencke T. The influence of residual neuromuscular block on the incidence of critical respiratory events. A randomised, prospective, placebo-controlled trial. Eur J Anaesthesiol. 2011 Dec;28(12):842-8. doi: 10.1097/EJA.0b013e328345cd11. PMID 21455074